CLINICAL TRIAL: NCT03010943
Title: Chirurgie Eveillee du Cerveau Sous Realite Virtuelle Integree Aux Outils Bloc Operatoire : Etude de Tolerance
Brief Title: Brain Awake Surgery Using Virtual Reality Headset
Acronym: CERVO1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A01139-42
Record Dates: First submitted 2016-12-15; First posted 2017-01-05 (Estimated); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Brain Tumor; Virtual Reality
Keywords: virtual reality; glioma surgery; awake craniotomy; brain tumor; glioma; neurosurgery
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain surgery with virtual reality headset (Experimental)
  Interventions: Device: Virtual reality headset

INTERVENTIONS:
Device: Virtual reality headset — Feasibility and tolerance
  Other Names: awake craniotomy

SUMMARY:
Feasibility and tolerance study of virtual reality headset for brain mapping during brain awake surgery.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral tumor or any type of brain lesion localized at the vicinity of eloquent area

Exclusion Criteria:

* Emergency
* Any contra-indication to awake brain surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
percentage of patients in which assessment of language functions during awake craniotomy, is possible with virtual reality headset. | During awake surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MENEI, MDPHD, Study Director — University hospital of Angers
Locations (1):
- CHU Angers, Angers, France

REFERENCES:
- [Result] Mazerand E, Le Renard M, Hue S, Lemee JM, Klinger E, Menei P. Intraoperative Subcortical Electrical Mapping of the Optic Tract in Awake Surgery Using a Virtual Reality Headset. World Neurosurg. 2017 Jan;97:424-430. doi: 10.1016/j.wneu.2016.10.031. Epub 2016 Oct 15. PMID 27756671
- [Derived] Casanova M, Clavreul A, Soulard G, Delion M, Aubin G, Ter Minassian A, Seguier R, Menei P. Immersive Virtual Reality and Ocular Tracking for Brain Mapping During Awake Surgery: Prospective Evaluation Study. J Med Internet Res. 2021 Mar 24;23(3):e24373. doi: 10.2196/24373. PMID 33759794
- [Derived] Bernard F, Lemee JM, Aubin G, Ter Minassian A, Menei P. Using a Virtual Reality Social Network During Awake Craniotomy to Map Social Cognition: Prospective Trial. J Med Internet Res. 2018 Jun 26;20(6):e10332. doi: 10.2196/10332. PMID 29945859